CLINICAL TRIAL: NCT01836341
Title: A Dose-Finding Study Of Afatinib In Combination With Cisplatin Or Carboplatin + Pemetrexed In Patients With EGFR-Mutant Lung Cancers Undergoing Definitive Chemoradiation
Brief Title: Afatinib In Combination With Cisplatin Or Carboplatin + Pemetrexed In Patients With EGFR-Mutant Lung Cancers Undergoing Definitive Chemoradiation
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Boehringer Ingelheim (Industry); National Comprehensive Cancer Network (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-279
Record Dates: First submitted 2013-04-17; First posted 2013-04-19 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2013-12

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Afatinib; Cisplatin; Carboplatin; Pemetrexed; Radiation therapy; EGFR mutation; 12-279
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Afatinib; Cisplatin; Carboplatin; Pemetrexed; Radiotherapy

ARMS (1):
- Afatinib w Cisplatin Pemetrexed Chemoradiation (Experimental): induction afatinib 40mg daily x 28days Cisplatin or Carboplatin (can be used if patient is not eligible for cisplatin) + Pemetrexed + 50Gy to pretreatment field boost to 60Gy to residual tumor + afatinib dose escalation*
  *afatinib dose levels: 20mg daily, 30mg daily & 40mg daily (3+3 design) Then adjuvant afatinib x 2 years
  Interventions: Drug: Afatinib; Drug: Cisplatin; Drug: Carboplatin; Drug: Pemetrexed; Radiation: Radiation therapy

INTERVENTIONS:
Drug: Afatinib
Drug: Cisplatin
Drug: Carboplatin
Drug: Pemetrexed
Radiation: Radiation therapy

SUMMARY:
The purpose of this Phase I study is to test the safety of combining afatinib with standard chemotherapy and radiation. The drug afatinib will be given before the chemotherapy and radiation therapy to shrink the tumor and evaluate how afatinib affects the patient. This study will then test the safety of afatinib at different dose levels when combined with the chemotherapy drugs cisplatin or carboplatin, and pemetrexed. These treatments will be given during radiation treatment and the drug afatinib will be continued after chemotherapy and radiation.

ELIGIBILITY:
Inclusion Criteria:

* Unresectable or inoperable, stage III or locoregional recurrence without evidence of distant, metastatic disease
* Pathologic confirmation of NSCLC at MSKCC
* Documentation of a sensitizing EGFR mutation
* Age ≥ 18 years
* No contraindication to definitive thoracic radiation therapy with concurrent chemotherapy

Adequate organ function as defined by:

* Calculated creatinine clearance≥ 45 mL/min (by Cockcroft-Gault)
* Total bilirubin less than 1.5 x ULN (unless known Gilbert's disease) and AST/ALT less than 3 x ULN
* Absolute neutrophil count greater than 1500/mm3
* Platelet count greater than 100,000/mm3
* Women of childbearing age must have a negative blood pregnancy test
* Men and women of childbearing potential must be willing to use effective contraception while on treatment and for at least 3 months there after

Exclusion Criteria:

* Prior chemotherapy or radiation therapy for this lung cancer (history of prior lung cancer that has been treated and deeded inactive by the clinician is acceptable)
* Ineligible for cisplatin or carboplatin per medical oncologist
* Ineligible for pemetrexed per medical oncologist
* Greater than minimal, exudative, or malignant pleural effusion
* Calculated creatinine clearance by Cockcroft & Gault method ≤45 ml/min
* Unstable congestive heart failure
* Ejection fraction <50% as assessed by MUGA or echocardiogram
* Interstitial lung disease
* Patient requiring on-going treatment with a potent inhibitor (cyclosporin, erythromycin, ketoconazole, itraconazole, quinidine, phenobarbital with quinidine, ritonavir, valspodar, verapamil) or inducer of P-gp (St. John's wort or rifampin)
* Women who are breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-04; Primary Completion 2015-04 (Estimated); Study Completion 2015-04 (Estimated)

PRIMARY OUTCOMES:
maximum tolerated dose | 1 year
  This will be defined as the dose at which fewer than 1:6 patients experiences a dose-limiting toxicity.

SECONDARY OUTCOMES:
local control rate | at 1 year and at 2 years
  will be determined as the proportion of patients who start the concurrent phase who are alive and free of local failure.
tolerability of adjuvant afatinib | at 3 months
  Tolerability will be defined by in terms of dose reductions, delays and discontinuations of patients who have not had disease progression or death.
median progression free survival | 2 years
  PFS is defined as the duration of time from start of treatment to time of progression of disease or death, whichever occurs first.
median overall survival | 2 years
  will be calculated using Kaplan-Meier estimates among all patients enrolled.

CONTACTS AND LOCATIONS:
Overall Officials: Jamie E. Chaft, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org/